CLINICAL TRIAL: NCT02277119
Title: Topcon 3D OCT-1 Maestro Optic Disc and RNFL Study: Agreement and Repeatability Comparison With the iVue
Brief Title: Clinical Study of the Optic Disc Parameters
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Topcon Medical Systems, Inc. (Industry)
Responsible Party: Sponsor
Organization: Topcon Corporation (Industry)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: Maestro2
Record Dates: First submitted 2014-10-21; First posted 2014-10-28 (Estimated); Results first posted 2016-11-02 (Estimated); Last update posted 2022-06-28 (Actual); Status verified 2022-06

CONDITIONS: Normal Healthy Subjects With No Known Ocular Diseases; Glaucomatous Eyes; Eyes With Retinal Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Normal Eyes (Experimental): Subjects with no known ocular diseases will be scanned with the iVue and Maestro device
  Interventions: Device: Maestro; Device: iVue
- Glaucomatous Eyes (Experimental): Subjects presenting with different stages of glaucoma will be scanned with the iVue and Maestro device
  Interventions: Device: Maestro; Device: iVue
- Eyes with Retinal Diseases (Experimental): Subjects presenting with Retinal pathological eyes will be scanned on the iVue and Maestro device
  Interventions: Device: Maestro; Device: iVue

INTERVENTIONS:
Device: Maestro — OCT machines used for diagnostic purposes
Device: iVue — OCT machines used for diagnostic purposes

SUMMARY:
Assess the repeatability and agreement of the Optic Disc Parameters, Retinal Nerve Fiber Layer (RNFL) Thickness, and Full Retinal Thickness between the Maestro and iVue OCT devices

ELIGIBILITY:
Inclusion Criteria for Normal Group

1. Subjects 18 years of age or older on the date of informed consent
2. Subjects able to understand the written informed consent and willing to participate as evidenced by signing the informed consent
3. Subjects presenting at the site with normal eyes (eyes without pathology)
4. lOPs 21mmHg bilaterally
5. BCVA 20/40 or better (each eye)
6. Both eyes must be free of eye disease

Exclusion Criteria for Normal Group

1. Subjects that have participated in any previous study using 3D OCT-1 Maestro device.
2. Subjects unable to tolerate ophthalmic imaging
3. Subject with ocular media not sufficiently clear to obtain acceptable OCT images
4. HFA visual field (24-2 Sita Standard, white on white) result abnormal, defined as GHT 'Outside Normal Limits' and/or PSD < 5%
5. HFA visual field (24-2 Sita Standard, white on white) result unreliable (based on manufacturer's recommendation), defined as fixation losses> 33% or false positives > 25%, or false negatives > 25%
6. Presence of any ocular pathology except for cataract
7. Previous ocular surgery or laser treatment, other than uncomplicated refractive procedure or cataract surgery, performed within six months prior to study scanning
8. Narrow angle
9. History of leukemia, dementia or multiple sclerosis
10. Concomitant use of hydroxychloroquine and chloroquine

Inclusion Criteria for Glaucoma Group

1. Subjects 18 years of age or older on the date of informed consent
2. Subjects able to understand the written informed consent and willing to participate as evidenced by signing the informed consent
3. Subjects presenting at the site with glaucoma
4. BCVA 20/40 or better in the study eye
5. HFA visual field (24-2 Sita Standard, white on white) result abnormal, defined as GHT 'Outside Normal Limits' and/or PSD < 5% in the study eye

Exclusion Criteria for Glaucoma Group

1. Subjects that have participated in any previous study using 3D OCT-1 Maestro device.
2. Subjects unable to tolerate ophthalmic imaging
3. Subject with ocular media not sufficiently clear to obtain acceptable OCT images
4. HFA visual field (24-2 Sita Standard, white on white) result unreliable, defined as fixation losses > 33% or false positives > 25%, or false negatives > 25% in the study eye
5. Presence of any ocular pathology except glaucoma in the study eye
6. Previous ocular surgery or laser treatment, other than uncomplicated refractive procedure or cataract surgery, performed within six months prior to study scanning in the study eye
7. History of leukemia, dementia or multiple sclerosis
8. Concomitant use of hydroxychloroquine and chloroquine

Inclusion Criteria for Retinal Group

1. Subjects 18 years of age or older on the date of informed consent
2. Subjects able to understand the written informed consent and willing to participate as evidenced by signing the informed consent
3. Subjects presenting at the site with retinal disease
4. lOP <= 21mmHg in the study eye
5. BCVA 20/400 or better in the study eye
6. Diagnosis of some type of retinal pathology by investigator, may include, but not limited to: Macular Degeneration, Diabetic Macular Edema, Diabetic Retinopathy, Macular Hole, Epiretinal Membrane, Cystoid Macula Edema, and others

Exclusion Criteria for Retinal Group

1. Subjects that have participated in any previous study using 3D OCT-1 Maestro device.
2. Subjects unable to tolerate ophthalmic imaging
3. Subject with ocular media not sufficiently clear to obtain acceptable OCT images
4. Presence of glaucoma or any ocular pathology other than a Retinal pathology (e.g., cornea pathology) in the study eye
5. Previous ocular surgery or laser treatment other than uncomplicated refractive procedure or cataract surgery performed within six months prior to study scanning in the study eye
6. Narrow angle in the study eye
7. History of leukemia, dementia or multiple sclerosis
8. Concomitant use of hydroxychloroquine and chloroquine

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2014-10; Primary Completion 2015-01 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mike Sinai, PhD, Study Director — Topcon Corporation
Locations (2):
- United States (2):
  - Western University of Health Sciences, Pomona, California
  - SUNY College of Optometry, New York, New York

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Normal Eyes | Glaucomatous Eyes | Eyes With Retinal Diseases
Started | 58 | 24 | 27
Completed | 55 | 20 | 19
Not Completed | 3 | 4 | 8
Not completed — Lack of Efficacy | 1 | 1 | 1
Not completed — Protocol Violation | 2 | 3 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Normal Eyes | Glaucomatous Eyes | Eyes With Retinal Diseases | Total
Number analyzed (Participants) | 58 | 24 | 27 | 109
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 55 | 16 | 19 | 90
  >=65 years | 3 | 8 | 8 | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.2 (13.3) | 57.8 (20.2) | 60.5 (13.4) | 48.7 (18.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 10 | 13 | 55
  Male | 26 | 14 | 14 | 54
Region of Enrollment [Number; unit: participants]
  United States | 58 | 24 | 27 | 109
Optic Disc Area Difference [Mean (Standard Deviation); unit: Microns Squared] | 0.197 (0.228) | 0.201 (0.262) | 0.097 (0.216) | 0.165 (0.235)

OUTCOME MEASURES:

1. Primary Outcome: Optic Disc Measurements (Optic Disc Size)
Description: Reporting of the Optic Disc Size difference between the Maestro and iVue
Time Frame: 1 Hour
Measure: Mean (Standard Deviation); unit: Mircrons squared
Arm/Group | Normal Eyes | Glaucomatous Eyes | Eyes With Retinal Diseases
Number analyzed (Participants) | 58 | 24 | 27
Mircrons squared | 0.197 (.228) | 0.097 (0.216) | 0.201 (0.262)

2. Primary Outcome: Retinal Nerve Fiber Layer (RNFL) Thickness Measurements
Description: RNFL thickness measured
Time Frame: 1 Hour
Measure: Mean (Standard Deviation); unit: Microns
Arm/Group | Normal Eyes | Glaucomatous Eyes | Eyes With Retinal Diseases
Number analyzed (Participants) | 58 | 24 | 27
Microns | 4.682 (4.333) | 2.526 (6.367) | 4.103 (8.789)

3. Primary Outcome: Full Retinal Thickness Measurement
Description: Full Retinal Thicknesses Measurement
Time Frame: 1 Hour
Population: Glaucomatous eyes were not scanned and analyzed in the Full Retina Thickness portion of the study. Since the imaging is done in a different area of the eye compare to Retinal Nerve Fiber Layer participants analyzed will be different between these measurement areas.
Measure: Mean (Standard Deviation); unit: Microns
Arm/Group | Normal Eyes | Glaucomatous Eyes | Eyes With Retinal Diseases
Number analyzed (Participants) | 19 | 0 | 18
Microns | 22.845 (11.482) |  | 21.299 (24.524)

4. Primary Outcome: Optic Disc Measurement (Cup Size)
Description: Reporting of the Cup size difference between the Maestro and iVue
Time Frame: 1 Hour
Measure: Mean (Standard Deviation); unit: Microns cubed
Arm/Group | Normal Eyes | Glaucomatous Eyes | Eyes With Retinal Diseases
Number analyzed (Participants) | 58 | 24 | 27
Microns cubed | 0 (0.072) | -0.003 (0.124) | 0.016 (0.065)

ADVERSE EVENTS:
Arm/Group | Normal Eyes | Glaucomatous Eyes | Eyes With Retinal Diseases
Serious Adverse Events (participants affected / at risk) | 0/58 | 0/24 | 0/27
Other Adverse Events (participants affected / at risk) | 0/58 | 0/24 | 0/27

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days